CLINICAL TRIAL: NCT04845477
Title: Effects of Magnetic Tape Over Hip Cutaneous Nerves in Patients With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francisco Selva (Other)
Responsible Party: Sponsor-Investigator, Francisco Selva, Principal Investigator, Clínica Dr. Francisco Selva
Organization: Clínica Dr. Francisco Selva (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23
Record Dates: First submitted 2021-04-08; First posted 2021-04-15 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Low Back Pain
Keywords: Magnetic tape; Range on motion; Cold; Cutaneous nerves; Hip; Kinovea® program
MeSH Terms: conditions — Low Back Pain; Common Cold

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- internal hip rotation pre measurement (No Intervention): with knee and hip flexion at 90º, internal hip rotation will be performed
- internal hip rotation post experimental application measurement (Experimental): with Magnetic tape Application with knee and hip flexion at 90º, internal hip rotation will be performed
  Interventions: Device: Magnetic tape
- internal hip rotation post placebo application measurement (Placebo Comparator): with Placebo tape Application with knee and hip flexion at 90º, internal hip rotation will be performed
  Interventions: Device: Kinesiology tape

INTERVENTIONS:
Device: Magnetic tape — magnetic tape is applied without creating any tension over the cutaneous nerves of the groin with less internal hip rotation
  Arms: internal hip rotation post experimental application measurement
Device: Kinesiology tape — kinesiology tape is applied without creating any tension over the cutaneous nerves of the groin with less internal hip rotation
  Arms: internal hip rotation post placebo application measurement

SUMMARY:
A tape is applied over the inguinal skin nerves in people with low back pain. When placing the experimental tape, mobility should be improved and when the area is cooled with the tape, rotation should be limited again by inhibiting skin receptors. When returning to the initial temperature, you should improve the degrees of mobility again demonstrating that Magnetic tape only acts on the dermal receptors.

The possible variation of the range in movement is measured with the validated program for the measurement of angles, Kinovea® program. A kinesiology tape was used as a placebo tape and the magnetic tape was used in a randomized experimental way.

DETAILED DESCRIPTION:
Detailed Description:

A double-blind randomized clinical trial is designed where subjects with low back pain will be selected and blinded to recieve the Magnetic Tape® or placebo Tape. Likewise, the evaluator who puts the Magnetic Tape® does not know what material he is using, as it is supplied by another researcher.

The recommendations of the "Consolidated Standards of Reporting Trials" (CONSORT) will be followed. All participants will receive a participant information sheet and sign informed consent. Patients aged 18 to 65 years with low back pain will be recruited from different private clinics in the city of Valencia, Spain.

The hypothesis is that when Magnetic Tape® comes into contact with electromagnetic fields such as those generated by living beings, due to the movement of electrical charges (ions), as defined by Ampere's Law, the domains of the tape are oriented or aligned in parallel with the external magnetic field creating a magnetic flux with a north pole and a south pole. This generated field in turn produces a magnetic induction proportional to the variation of the magnetic flux, as defined by the Faraday Law.

This electric potential produces a redistribution of the electric charge (ions) generating a magnetic field due to the orientation of the tape domains, then exerting a force on the moving charges within the electrolyte.

Physiological, Lorentz's Law, regulating Magnetic Tape® aberrant electromagnetic fields.

After signing the informed consent and data protection, the groups with low back pain will be formed that will receive the application of both Magnetic Tape® and the intervention of a placebo tape. To avoid that the order of the intervention influences the results of the study, the subjects will be randomized into two different groups, Group A and Group B. Group A will receive Magnetic tape® and Group B will do the opposite. The next day the other tape will be applied.

Passive joint ROM of both hips is assessed by placing the patient in a supine position with 90º hip and knee flexion, performing passive internal hip rotation. An infrared marker and the video camera are placed perpendicular to the hip joint so that when the lower limb is flexed, the knee coincides with that point so that the measurement is reproducible.

The infrared thermometer is placed on the subject at a height sufficient to frame the iliac fossa to be evaluated.

After recording the passive hip rotation maneuver, the joint ROM will be assessed using the Kinovea® program.

During the same movement, the muscle activation of the movement antagonist ipsilateral adductor longus will be assessed with the surface electromyograph so that it is not activated.

The local temperature variation of the ipsilateral iliac fossa will also be assessed with the infrared thermometer.

Subsequently, a 5-8 cm long by 5 cm wide strip of Magnetic Tape® will be placed over the ipsilateral iliac fossa of the hip with movement limitation to perform the passive internal rotation of the hip again and record the degrees of range of motion.

Next, the tape shall then be removed and a cold pack shall be placed on the skin. After reducing the local temperature, the cold pack shall be removed, the tape shall be reapplied and the passive internal rotation of the hip shall be measured.

The initial temperature shall be returned to the area and the passive internal rotation of the hip shall be recorded again with the tape.

Each subject shall be their own control as one tape shall be applied on one day and the other tape on the following test day.

Neither application has to be painful.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with low back pain.
* Subjects aged 18-65 years.

Exclusion Criteria:

* Tape allergies
* Adhesive allergies
* Pregnant
* People with pacemakers
* People who have any contraindication of electromagnetic fields
* People with neurological diseases
* Taking any medication that may interact with magnetic fields.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
range on motion | first assessment before placing the tapes. After placing one of the tape. After placing the other tape. After cooling the bandaged area with both tape. After recovery of local temperature.
  Maximum degrees of internal hip rotation measured with the Kinovea® program. Validated Video Program
Temperature | first evaluation before placing the tapes. After cooling the bandaged area with both tapes. After recovery of local temperature.
  an infrared thermometer will measure the temperature of the groin area in degrees centigrade

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Francisco Selva, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No